CLINICAL TRIAL: NCT04180436
Title: Pharmacokinetics and Pharmacodynamics of rivAroxaban After Bariatric Surgery and in mORBid Obesity
Brief Title: Pharmacokinetics of Rivaroxaban After Bariatric Surgery
Acronym: ABSORB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABSORB (29BRC19.0078)
Record Dates: First submitted 2019-07-19; First posted 2019-11-27 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2022-07

CONDITIONS: Bariatric Surgery; Morbid Obesity
Keywords: sleeve gastrectomy; gastric bypass; morbid obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- morbidly obese patients with BMI ≥ 40 (Experimental): Morbidly obese patients with BMI ≥ 40
  Interventions: Drug: rivaroxaban 20 mg once daily 8 days
- Patients operated by gastric bypass (Experimental): Patients operated by gastric bypass for over a year and with stable weight
  Interventions: Drug: rivaroxaban 20 mg once daily 8 days
- Patients operated by sleeve gastrectomy (Experimental): Patients operated by sleeve gastrectomy for over a year and with stable weight
  Interventions: Drug: rivaroxaban 20 mg once daily 8 days
- Control group: non-operated subjects (Experimental): Control group: non-operated subjects but with an age and a BMI corresponding to those of the patients of the 2 operated groups.
  Interventions: Drug: rivaroxaban 20 mg once daily 8 days

INTERVENTIONS:
Drug: rivaroxaban 20 mg once daily 8 days — Blood samples for the measurement of rivaroxaban PK parameters

SUMMARY:
Data on pharmacokinetics of rivaroxaban after bariatric surgery and in morbid obesity are sparse. The aim of this study is to assess the pharmacokinetic and pharmacodynamic parameters of rivaroxaban, used at a therapeutic anticoagulant dose, in patients with previous bariatric surgery, with sleeve gastrectomy or gastric bypass, and in morbid obese subjects.

Four groups of 16 subjects per group are studied: Morbid obese subjects / Subjects who have undergone gastric bypass surgery / Subjects who have undergone sleeve gastrectomy surgery / Non-operated control subjects matched for age and BMI with operated subjects.

All patients (obese, surgical patients, and controls) will receive rivaroxaban 20mg once daily during 8 days. Blood samples will be taken predose (Baseline) and 0.5, 1, 2, 3, 6, 9, 12 and 24h post rivaroxaban administration at day1 and day8. PK and PD parameters will be compared between groups in order to explore the impact of bariatric surgery, type of surgery and body mass index on the pharmacological profile of rivaroxaban.

ELIGIBILITY:
Inclusion Criteria:

* Creatinine clearance measured by the Cockroft formula ≥ 60 mL / min
* Patient meeting the specific criteria of one of the 4 groups:
* morbidly obese patients with BMI ≥ 40
* Patients operated by gastric bypass for over a year and with stable weight
* Patients operated by sleeve gastrectomy for over a year and with stable weight
* Control group: non-operated subjects but with an age and a BMI corresponding to those of the patients of the 2 operated groups.

Exclusion Criteria:

* Indication for anticoagulant therapy, antiplatelet therapy or long-term nonsteroidal anti-inflammatory drugs
* Clinically significant bleeding in progress
* Taking oral or parenteral anticoagulants, or taking platelet antiaggregants within 4 weeks before inclusion
* Congenital or acquired hemorrhagic disorders (eg von Willebrand disease, hemophilia)
* Injury or disease, at significant risk of major bleeding (gastrointestinal ulceration, presence of malignant tumors with a high risk of bleeding, recent brain or spinal cord injury, recent cerebral, spinal or ophthalmic surgery, recent intracranial hemorrhage, known or suspected oesophageal varices , arteriovenous malformations, vascular aneurysms or major intraspinal or intracerebral vascular abnormalities)
* Severe uncontrolled arterial hypertension
* Active gastrointestinal disease potentially leading to bleeding disorders (esophagitis, gastritis, gastroesophageal reflux disease, chronic inflammatory bowel disease)
* Vascular retinopathy
* Bronchiectasis or history of pulmonary bleeding
* Hypersensitivity to the active substance or to any of the excipients of rivaroxaban
* Hepatic involvement associated with coagulopathy and clinically significant bleeding risk, including cirrhotic patients with Child Pugh Grade B or C score
* Concomitant use of potent inhibitors or inducers of CYP3A4 and / or P-gp (azole antifungal or HIV protease inhibitor)
* Participation in a paid and / or therapeutic study in the previous 3 months
* Pregnant or lactating women,
* Women of childbearing potential not using effective contraception

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
AUC of rivaroxaban | up to 8 days
  Rivaroxaban plasma concentrations was assessed by the reference method at the different sampling points to determine the area under the curve (AUC)
Cmax of rivaroxaban | up to 8 days
  Cmax of rivaroxaban was assessed
Tmax of rivaroxaban | up to 8 days
  Tmax of rivaroxaban was assessed

SECONDARY OUTCOMES:
Prothrombin time | up to 8 days
  Prothrombin time of rivaroxaban was assessed
Activated partial thromboplatin time (aPTT) | up to 8 days
  Activated partial thromboplatin time was assessed
Fibrinogen levels | up to 8 days
  Fibrinogen levels was was assessed
Rivaroxaban anti-Xa activity | up to 8 days
  Rivaroxaban anti-Xa activity was assessed
Rate of bleedings | up to 15 days
  Treatment-Related Adverse Events were assessed
Other adverse events | up to 15 days
  Number of other adverse events than bleedings was assessed
Thrombin generation test of rivaroxaban | up to 8 days
  Thrombogram (thrombin generation test) data for each time analyzed allows measurement of peak height . These data will be used to model the PD of rivaroxaban and to estimate the PD variability.
Thrombin generation test of rivaroxaban | up to 8 days
  Thrombogram (thrombin generation test) data for each time analyzed allows measurement of thrombin generation potential (FTE). These data will be used to model the PD of rivaroxaban and to estimate the PD variability.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Result] Leven C, Delavenne X, Roche C, Bressollette L, Couturaud F, Lacut K, Thereaux J. Full-dose rivaroxaban in patients with a history of bariatric surgery: bridging the knowledge gap through a phase 1 study. J Thromb Haemost. 2024 Oct;22(10):2844-2854. doi: 10.1016/j.jtha.2024.06.024. Epub 2024 Jul 11. PMID 39002729